CLINICAL TRIAL: NCT06687447
Title: The Effect of Oxytocin Massage and Reflexology Applied to Primiparous Mothers After Cesarean Section on Insufficient Milk Perception, Breastfeeding Motivation, Fatigue, Anxiety and Uterus Involution
Brief Title: The Effect of Two Methods Applied to Mothers on Insufficient Milk Perception, Breastfeeding Motivation, Fatigue, Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Büşra Nur GELDİ, Nurse, PhD Student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ODU-HSI-BNG-01
Record Dates: First submitted 2023-12-28; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Caesarean Section
Keywords: reflexology; oxytocin massage; fatigue; anxiety; milk production
MeSH Terms: conditions — Fatigue; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It was planned for three groups: oxytocin massage group, reflexology group and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Random distribution of women included in the study to intervention groups and control groups was carried out at www.random.org. Which groups were intervention or control groups were determined by drawing lots at the beginning of the study. The numbers in the intervention groups and the control group will be placed in opaque envelopes, and the group in which the women who meet the criteria will be will be decided by drawing lots of sealed envelopes after the pre-test data is completed.The statistical analysis phase is blind since an independent statistician other than the researcher will perform the statistical analysis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oxycotin Massage Group (Active Comparator): The researcher will perform oxytocin massage to the fifth-sixth rib along the patient's spine.
  Interventions: Other: Oxycotin Massage Group
- Reflexology Group (Active Comparator): The researcher will apply pressure in different ways to the reflex points on the patient's sole with her fingers.
  Interventions: Other: Reflexology Group
- Control Group (Other): Patients in the control group will not undergo any intervention and will receive their routine care.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Oxycotin Massage Group — Primiparous women will be visited 12 hours after cesarean delivery, women will be informed, verbal and written consent will be obtained from women who want to participate in the study, and pre-test data will be collected by the researcher. The pre-test data of the research were it will be collected by face-to-face interview technique in approximately 25 minutes. The height of the fundus part of the uterus will be measured with a tape measure. The woman's physiological parameters will be measured by the researcher. At this stage, the patient will receive an oxytocin massage for 10 minutes while in a sitting position. One hour after the application (13th hour after cesarean section), the physiological parameters of the patients will be measured again by the researcher. 24 hours after the application (36 hours after cesarean section), the data of the patients will be collected again by the researcher and uterine involution and physiological parameters will be evaluated.
  Arms: Oxycotin Massage Group
Other: Reflexology Group — Primiparous women will be visited 12 hours after cesarean delivery, women will be informed women who want to participate in the study, and pre-test data will be collected. The pre-test data of the research were it will be collectedapproximately 25 minutes. The height of the fundus part of the uterus will be measured with a tape measure. The woman's physiological parameters will be measured. In practice; The foot is first relaxed and warmed up with passive movements, then the sole of the foot is scanned with the thumb walking crawling technique. The application will be applied first to the right foot for 10 minutes and then to the left foot for a total of 20 minutes. One hour after the application (13th hour after cesarean section), the physiological parameters of the patients will be measured again. 24 hours after the application (36 hours after cesarean section), the data of the patients will be collected again and uterine involution and physiological parameters will be evaluated.
  Arms: Reflexology Group
Other: Control Group — Primiparous women will be visited 12 hours after cesarean delivery, women will be informed, verbal and written consent will be obtained from women who want to participate in the study, and pre-test data will be collected by the researcher. The pre-test data of the research were it will be collected by face-to-face interview technique in approximately 25 minutes. The height of the fundus part of the uterus will be measured with a tape measure. The woman's physiological parameters will be measured by the researcher. Patients in the control group will not undergo any intervention and will receive their routine care. One hour after the application (13th hour after cesarean section), the physiological parameters of the patients will be measured again by the researcher. 24 hours after the application (36 hours after cesarean section), the data of the patients will be collected again by the researcher and uterine involution and physiological parameters will be evaluated.
  Arms: Control Group

SUMMARY:
Although the World Health Organization predicts the caesarean section rate to be 10-15%, the caesarean section rate in Turkey is 52%, more than three times the international standard. It is very important to eliminate the physical and psychosocial problems experienced by women during this period, to encourage breastfeeding, and at the same time to protect and improve maternal health. Maintaining the mother's well-being after cesarean section and supporting pharmacological treatment with non-pharmacological practices have an important place in nursing care. Therefore, this study will examine the effects of oxytocin massage and reflexology applied to mothers in the post-cesarean period on the perception of insufficient milk, breastfeeding motivation, fatigue, anxiety and uterine involution.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who gave birth at the age of 18 and over
* The one who is married
* At least primary school graduate,
* Primiparous mothers who gave birth by cesarean section,
* Having a single, healthy newborn at full term,
* Those who did not experience any problems during pregnancy and the early postpartum period,
* The tissue integrity in the area to be applied is complete and healthy,
* Breastfeeding her baby after birth,
* The baby is healthy, has no problems with the sucking reflex and does not have any congenital anomalies,
* Women who agree to participate in the research will be included in the study.

Exclusion Criteria:

* Those who gave birth by cesarean section before the 37th week of pregnancy,
* Women who gave birth by cesarean section with combined anesthesia,
* Discharged before 36 hours after birth,
* Having chronic diseases such as heart disease, diabetes, hypertension,
* Those with infectious diseases, infections, open wounds, masses, fractures, dislocations, deformities, varicose veins, burns, eczema, hematomas, thrombophlebitis, deep vein thrombosis on the foot skin,
* Experiencing any postpartum complications,
* Their baby is not with their mother for any reason,
* Those who have received a psychiatric diagnosis such as anxiety and depression,
* Women who want to leave the research at any stage of the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-06 (Estimated)

PRIMARY OUTCOMES:
Insufficient Milk Perception Scale | 36 hours
  The Insufficient Milk Perception Scale consists of a total of 6 questions and a single subscale. The first question on the scale is whether the mother finds her milk sufficient. The first question is answered as yes or no. The other 5 questions are scored between 0-10. The given score indicates that as it approaches zero, the mother perceives her milk as inadequate, and as she approaches 10, she perceives enough. A minimum of zero points and a maximum of 50 points can be obtained from the scale. The high score indicates that milk is sufficiently perceived.
Primipar Breastfeeding Motivation Scale | 36 hours
  The Insufficient Milk Perception Scale consists of a total of 6 questions and a single subscale. The first question on the scale is whether the mother finds her milk sufficient. The first question is answered as yes or no. The other 5 questions are scored between 0-10. The given score indicates that as it approaches zero, the mother perceives her milk as inadequate, and as she approaches 10, she perceives enough. A minimum of zero points and a maximum of 50 points can be obtained from the scale. The high score indicates that milk is sufficiently perceived.
Visual Similarity Scale for Fatigue (VAS-F) | 36 hours
  The scale consists of 29 items and has a 7-point Likert type and 4 sub-dimensions. These sub-dimensions; the value given to breastfeeding (items 1,2,4,6,8,10,12,14,15,20,24,25,28), self-efficacy (items 9,16,17,18,19,26,29 ), midwife support (items 21,22,23,27), success expectation (items 3,5,7,11,13). As the score obtained from each sub-dimension increases, the breastfeeding motivation level of that sub-dimension increases.
The State-Trait Anxiety Inventory (STAI) | 36 hours
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. It also is often used in research as an indicator of caregiver distress. Form has 20 items for assessing for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.

SECONDARY OUTCOMES:
Uterine Involution Evaluation Form | 36 hours
  This form is a form prepared by the researcher in line with the literature, in which the measurement of the length of the uterus is recorded and the uterine involution process of postpartum women is evaluated. The length of the uterus; It will be done by measuring the distance between the fundus of the uterus and the symphysis pubis with the help of a tape measure. When measuring uterine length, women will be ensured that their bladder is empty and the same tape measure will be used in all measurements.
Physiological Parameters Evaluation Form | 36 hours
  In this study, heart rate, body temperature, oxygen saturation, respiratory rate and blood pressure values will be measured and recorded in the Physiological Parameters Form.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Nur GELDİ, Principal Investigator — Ordu University; Nülüfer ERBİL, Study Director — Ordu University
Locations (1):
- Büşra Nur GELDİ, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No